CLINICAL TRIAL: NCT00611650
Title: Phase II Trial of Polyphenon E in Current and Former Smokers With Bronchial Dysplasia
Brief Title: Green Tea Extract in Treating Current or Former Smokers With Bronchial Dysplasia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000578224; P01CA096964 (NIH); BCCA-H07-02401; H07-02401
Record Dates: First submitted 2008-02-08; First posted 2008-02-11 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer; Precancerous Condition; Tobacco Use Disorder
Keywords: non-small cell lung cancer; squamous lung dysplasia; tobacco use disorder
MeSH Terms: conditions — Lung Neoplasms; Precancerous Conditions; Tobacco Use Disorder; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral Polyphenon E twice daily for 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: defined green tea catechin extract
- Arm II (Placebo Comparator): Patients receive a placebo twice daily for 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: defined green tea catechin extract — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. The use of Polyphenon E, a substance found in green tea, may keep cancer from forming in current or former smokers with bronchial dysplasia.

PURPOSE: This randomized phase II trial is studying the side effects and how well green tea extract works in treating current or former smokers with bronchial dysplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy and safety of Polyphenon E, a defined green tea catechin extract, in current or former smokers with bronchial dysplasia and increased inflammatory load as measured by C-reactive protein.

Secondary

* To evaluate the ability of Polyphenon E to modulate other surrogate endpoint biomarkers of oxidation stress, inflammation, aberrant methylation, cell cycle regulation, apoptosis, oncogene/tumor suppressor gene expression, as well as phase I and II enzyme regulation in biological samples from these patients.
* To establish a library of optical coherent tomography (OCT) images of the bronchial epithelium with corresponding histopathology, nuclear morphometry, and other biomarker information.
* To assess the potential of OCT as a non-biopsy method for evaluating chemoprevention agents.

OUTLINE: This is a multicenter study. Patients are stratified by gender. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral Polyphenon E twice daily for 3 months in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive a placebo twice daily for 3 months in the absence of disease progression or unacceptable toxicity.

Patients undergo standard white-light bronchoscopy and fluorescence bronchoscopy with optical coherence tomography (OCT) at baseline and at 3 months. During these procedures, patients are evaluated using the Onco-LIFE clinical device, which digitally records OCT images of abnormal areas or areas suspicious for intraepithelial neoplasia or invasive carcinoma. Once these areas have been localized, patients are biopsied under fluorescence bronchoscopy guidance to obtain both dysplastic bronchial epithelial tissue and normal bronchial mucosa. Biopsy specimens are examined by immunostaining for tissue-based biomarkers (i.e., Ki-67, cleaved caspase-3, p53, and VEGF). Patients also undergo oral brushing, bronchial brushing, and bronchoalveolar lavage at baseline and at 3 months to obtain bronchial epithelial cells for differential gene expression and methylation biomarker studies (e.g., cDNA microarray analysis, polymerase chain reaction, and northern blotting). Cytokines and other molecular biomarkers (i.e., C-reactive protein, surfactant protein D, oxidized glutathione, interleukin [IL]-6, IL-13, and macrophage inflammatory protein-1 levels) are measured in blood and bronchoalveolar lavage fluid samples by enzyme-linked immunoassay. Plasma EGCG levels are assessed by high-performance liquid chromatography. Urine cotinine levels and exhaled carbon monoxide levels are also assessed.

After completion of study therapy, patients are followed at 1 month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Current or former smoker who has smoked ≥ 30 pack-years (i.e., 1 pack per day for ≥ 30 years)

  * A former smoker is defined as one who has stopped smoking for ≥ 1 year
* C-reactive protein level > 1.2 mg/L
* One or more areas of dysplasia with a surface diameter > 1.2 mm on autofluorescence bronchoscopy
* No carcinoma in situ or invasive cancer on bronchoscopy
* No abnormal spiral chest CT scan suspicious of lung cancer

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Willing to take Polyphenon E or placebo twice a day regularly
* Willing to undergo bronchoscopy and spiral chest CT scan
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Creatinine normal
* Bilirubin normal
* AST and ALT normal
* Alkaline phosphatase normal
* No chronic active hepatitis or liver cirrhosis
* No severe heart disease (e.g., unstable angina or chronic congestive heart failure)
* No ongoing gastric ulcer
* No acute bronchitis or pneumonia within the past month
* No known reaction to xylocaine, salbutamol, midazolam, or alfentanil
* No known allergy to green tea and/or corn starch, gelatin, or other nonmedicinal ingredients
* No medical condition, such as acute or chronic respiratory failure or bleeding disorder, that, in the opinion of the investigator, could jeopardize patient safety during study participation

PRIOR CONCURRENT THERAPY:

* No concurrent consumption of > 7 cups of tea a week
* No other concurrent natural health products containing green tea compounds
* No concurrent antiarrhythmic agents
* No concurrent anticoagulants, such as warfarin or heparin

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-10; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in the severity of dysplasia (as defined by WHO criteria) in bronchial biopsy specimens as assessed at baseline and at 3 months | 3 months

SECONDARY OUTCOMES:
Change in the morphometric index in bronchial biopsy specimens as assessed at baseline and at 3 months | 3 months
Change in the concentrations (or grades) of Ki-67, p53, cleaved caspase-3, and VEGF in bronchial biopsy specimens as assessed by immunostaining at baseline and at 3 months | 3 months
Methylation biomarkers in bronchoalveolar lavage (BAL) cells as assessed at baseline and at 3 months | 3 months
Oncogene/ tumor suppressor gene expression in bronchial brush cells as assessed by cDNA microarray analysis at baseline and at 3 months | 3 months
Phase I and II enzyme regulation in bronchial brush cells as assessed by Affymetrix microarray analysis at baseline and at 3 months | 3 months
Change in C-reactive protein levels in plasma as assessed by enzyme-linked immunoassay (ELISA) at baseline and then monthly for 3 months | 3 months
Volumetric measurement of CT-detected lung nodules at baseline and then every 3-12 months for up to 24 months, depending on the size of the nodule | 24 months
Change in the concentrations (or grades) of surfactant protein D, oxidized glutathione, interleukin (IL)-6, IL-13, and MPIF-1 in plasma and BAL cells as assessed by ELISA at baseline and at 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lam, MD, Study Chair — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia, Canada